CLINICAL TRIAL: NCT06166615
Title: The Safety and Efficacy of 5-HT3 Receptor Antagonist (Ramosetron) Versus Psyllium (Agio®) for the Treatment of Fecal Incontinence: Multicenter Randomized Trial (SERAFI)
Brief Title: The Safety and Efficacy of 5-HT3 Receptor Antagonist (Ramosetron) for the Treatment of Fecal Incontinence
Acronym: SERAFI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Rumi Shin, Associate Professor of Medicine, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2303-158-1417
Record Dates: First submitted 2023-10-29; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — ramosetron; Psyllium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyllium group (Active Comparator): Take 2 sachets (12 g) orally once daily. Increase or decrease the dose as needed to treat your symptoms, with a maximum daily dose of 18 grams (6 grams in the morning and 12 grams in the evening). Do not chew this medication and take it with 1 to 2 cups of water.
  Take it for 1 month
  Interventions: Drug: Psyllium
- Ramosetron group (Experimental): Men: 5 μg orally once daily. Increase or decrease the dose as needed based on symptoms, with a minimum daily dose of 2.5 μg and a maximum daily dose of 10 μg.
  Women: 2.5 μg orally once daily. Women: 2.5 μg orally once daily, titrated up or down as needed, with a maximum daily dose of 5 μg.
  Take it for 1 month
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ramosetron — Ramosetron (a 5-HT3 receptor antagonist) has been developed as an effective treatment for irritable bowel syndrome-diarrhea (IBD-D) and is used to decrease intestinal motility, stiffen stool consistency, and reduce the number of urgency bowel movements. Since one of the goals of treatment for fecal incontinence is the maintenance of stool consistency, this agent is expected to be effective in treating fecal incontinence.
  Arms: Ramosetron group
Drug: Psyllium — Psyllium was found to be the most effective at improving symptoms of fecal incontinence among several dietary fibers in a randomized, controlled, single-blind study and is currently used as a first-line treatment for fecal incontinence.
  Arms: Pyllium group

SUMMARY:
This clinical trial aims to assess the effectiveness of Ramosetron compared to Psyllium, a gold standard therapy, in patients with fecal incontinence. The primary questions it seeks to answer are:

1. Does Ramosetron improve the symptoms of fecal incontinence?
2. Is Ramosetron superior to Psyllium in terms of symptom improvement and its impact on quality of life?

Participants will be randomly assigned to one of two groups, either taking Ramosetron or Psyllium for one month. They will be asked to complete a questionnaire. Researchers will then compare the Fecal Incontinence Severity Index between the Ramosetron and Psyllium groups to determine whether Ramosetron provides superior symptom relief compared to Psyllium.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with fecal incontinence (patients with 2 or more symptoms of fecal incontinence per month for at least 3 months).
2. Patients who are able to understand and comply with this study.
3. Individuals who are agreeable to being on contraception for the duration of the study.

Exclusion Criteria:

1. Patients who have difficulty swallowing medications
2. Patients with gastrointestinal deformities due to surgery
3. Patients with malabsorption
4. Patients with inflammatory bowel disease (IBD)
5. Patients undergoing treatment for cancer of the gastrointestinal tract
6. Patients who are allergic to the study drug
7. Patients with overflow incontinence and fecal impaction on rectal residual examination (DRE) or Bristol Stool Scale of 3 or less.
8. Patients taking medication for fecal incontinence within 1 month of study entry.
9. Pregnant or lactating women.
10. Patients with contraindications to any of the study drugs (i.e., intestinal obstruction, intestinal stones, acute abdomen, undiagnosed abdominal pain/nausea/vomiting, gastrointestinal stenosis and dysphagia, patients with megacolon syndrome, severe diabetes, etc.).
11. Patients taking an agent that is contraindicated in combination with either study drug.
12. Patients deemed by the investigator and staff to be unsuitable for participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference of Fecal Incontinence Severity Index | The FISI scores will be assessed at two time points - at baseline (prior to the initiation of treatment) and at 1 month post-treatment initiation.
  This outcome measure assesses the difference in Fecal Incontinence Severity Index (FISI) scores in patients with fecal incontinence before and after treatment. The FISI questionnaire, used in previous studies, will be utilized to compare the scores pre- and post-medication for both the Ramosetron group and the Psyllium Agio® group.
  Details about the FISI Scale:
  Unabbreviated Scale Title: Fecal Incontinence Severity Index (FISI) Scale Range: The FISI scale typically ranges from 0 to a maximum value 61. Interpretation of Scores: Higher scores on the FISI scale indicate a worse outcome, reflecting greater severity of fecal incontinence symptoms.

SECONDARY OUTCOMES:
Difference in Fecal Incontinence Severity Index (FISI) Scores Between the Two Groups | Measured at baseline and 1-,4-, and 12-month.
  This measure will assess the difference in FISI scores between the two treatment arms (Ramosetron group vs. Psyllium Agio® group).
  FISI Scale Details:
  Unabbreviated Scale Title: Fecal Incontinence Severity Index (FISI) Scale Range: 0-61 Score Interpretation: Higher FISI scores indicate worse fecal incontinence severity.
Fecal Incontinence Quality of Life Scale (FIQL) Scores Comparison | Measured at baseline and 1-,4-, and 12-month.
  This outcome measure assesses the impact of fecal incontinence on patients' quality of life using the FIQL. The FIQL is a patient-reported outcome measure (PROM) that evaluates four domains of quality of life: lifestyle, coping/behavior, depression/self-perception, and embarrassment. It consists of 4 questions and 29 items, with various response categories and scoring methods.
  Scale Range: The FIQL does not provide an overall score, which complicates its use and interpretation.The FIQL includes a range of response options across its items, from 1 to 4 for most items, 1 to 5 for one item, and 1 to 6 for another. Lower scores indicate lower quality of life.
  Score Interpretation: Higher scores in specific domains (e.g., depression/self-perception) may indicate worse outcomes in those areas.
Bristol Stool Scale Scores Comparison | Measured at baseline and 1-,4-, and 12-month.
  This measure will compare the Bristol Stool Scale scores between the two groups.
  Bristol Stool Scale Details:
  Unabbreviated Scale Title: Bristol Stool Scale Scale Range: 1-7 Score Interpretation: The scale classifies the form of human feces into seven categories.

CONTACTS AND LOCATIONS:
Overall Officials: Rumi Shin, MD, PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scarlett Y. Medical management of fecal incontinence. Gastroenterology. 2004 Jan;126(1 Suppl 1):S55-63. doi: 10.1053/j.gastro.2003.10.007. PMID 14978639
- [Background] Wald A, Bharucha AE, Cosman BC, Whitehead WE. ACG clinical guideline: management of benign anorectal disorders. Am J Gastroenterol. 2014 Aug;109(8):1141-57; (Quiz) 1058. doi: 10.1038/ajg.2014.190. Epub 2014 Jul 15. PMID 25022811
- [Background] Omar MI, Alexander CE. Drug treatment for faecal incontinence in adults. Cochrane Database Syst Rev. 2013 Jun 11;2013(6):CD002116. doi: 10.1002/14651858.CD002116.pub2. PMID 23757096
- [Result] Markland AD, Burgio KL, Whitehead WE, Richter HE, Wilcox CM, Redden DT, Beasley TM, Goode PS. Loperamide Versus Psyllium Fiber for Treatment of Fecal Incontinence: The Fecal Incontinence Prescription (Rx) Management (FIRM) Randomized Clinical Trial. Dis Colon Rectum. 2015 Oct;58(10):983-93. doi: 10.1097/DCR.0000000000000442. PMID 26347971
- [Result] Ryoo SB, Park JW, Lee DW, Lee MA, Kwon YH, Kim MJ, Moon SH, Jeong SY, Park KJ. Anterior resection syndrome: a randomized clinical trial of a 5-HT3 receptor antagonist (ramosetron) in male patients with rectal cancer. Br J Surg. 2021 Jun 22;108(6):644-651. doi: 10.1093/bjs/znab071. PMID 33982068
- [Derived] Park J, Ahn HM, Ryoo SB, Oh Y, Choi JS, Oh HK, Shin R. The Safety and Efficacy of Ramosetron versus Psyllium for the Treatment of Fecal Incontinence (SERAFI): Study protocol for a randomized, parallel, non-inferiority trial. Trials. 2025 Nov 5;26(1):471. doi: 10.1186/s13063-025-09165-2. PMID 41194155